CLINICAL TRIAL: NCT00837031
Title: A Phase II Study of Lenalidomide in Combination With Gemcitabine in Subjects With Untreated Advanced Carcinoma of the Pancreas
Brief Title: Lenalidomide With Gemcitabine in Treatment of Untreated Advanced Carcinoma of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 106
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic; Pancreatic Cancer; Lenalidomide; Revlimid; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Lenalidomide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): The study began with a lead-in portion to confirm the tolerability of lenalidomide (25mg PO days 1-21) in combination with gemcitabine (1000mg/m2 IV days 1, 8, and 15).
  After completion of the lead-in phase, all subsequent patients received lenalidomide 25mg PO on days 1-21 and gemcitabine 1000mg/m2 IV days 1, 8, and 15 of 28-day treatment cycles. Patients were instructed to take lenalidomide at approximately the same time each morning. Patients were permitted to continue treatment until disease progression or intolerable toxicity occurred.
  Interventions: Drug: Lenalidomide; Drug: Gemcitabine

INTERVENTIONS:
Drug: Lenalidomide — The starting dose of lenalidomide for the lead-in portion will be 25 mg orally daily on Days 1-21, followed by a 7-day rest period (28-day cycle). If the 25-mg dose of lenalidomide is found to be intolerable or unsafe (i.e., if more than one of the 6 patients experience a DLT), then the dose will be reduced to 20 mg orally daily, and 6 additional patients will be treated. All patients will receive lenalidomide at the confirmed tolerable dose (either 25 mg or 20 mg given orally daily on Days 1-21 of a 28-day cycle) until disease progression. If the 20-mg daily dose is found to be intolerable or unsafe, enrollment will be put on hold.
  Other Names: Revlimid
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV will be administered on Days 1, 8, and 15 for a 28-day cycle.
  Other Names: Gemzar

SUMMARY:
To evaluate the 6-month overall survival, safety, and tolerability of lenalidomide in combination with standard gemcitabine as first-line treatment for patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Because the activity of lenalidomide addresses numerous mechanisms of carcinoma growth inhibition - including, but not limited to anti-angiogenesis - lenalidomide is being evaluated as part of induction chemotherapy regimens for solid tumors. This phase II study in previously untreated metastatic pancreatic cancer is designed to establish and test the appropriate lenalidomide dose and regimen in combination with gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign the informed consent form.
2. Patients >=18 years of age at the time of signing the informed consent form.
3. Ability to adhere to the study visit schedule and other protocol requirements.
4. Histological or cytological documentation of adenocarcinoma of the pancreas, with metastases not amenable to curative surgery or definitive radiation. Patients with locally advanced disease are not eligible.
5. Radiographic or clinical evidence of measurable advanced metastatic pancreatic carcinoma. Patients must have measurable disease according to the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) for target lesions.
6. Previous gemcitabine or 5-fluorouracil (5-FU) with radiation therapy as adjuvant therapy is permitted. Extended use of gemcitabine or 5-FU after completion of adjuvant radiation therapy is not permitted. No prior gemcitabine for metastatic disease or for primary treatment of locally advanced disease is allowed.
7. ECOG performance status of <=2 at study entry.
8. Laboratory test results within these ranges:

   * Absolute neutrophil count (ANC) ≥1,500 cells/mm3 (1.5 x 109/L)
   * Platelet count ≥100,000 cells/ mm3 (100 x 109/L)
   * Serum creatinine <=2.5 mg/dL
   * Total bilirubin <=2.0 mg/dL
   * AST (SGOT) and ALT (SGPT) <=3.0 x ULN or <=5 x ULN if hepatic metastases are present.
9. Prior history of malignancy (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast, or localized prostate cancer with PSA <1.0 ng/mL), unless the patient has been free of disease for >=3 years.
10. All study participants must be registered into the mandatory RevAssist® program, and must be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

1. Prior use of systemic therapy for the treatment of adenocarcinoma of the pancreas, with the exception of 5-fluorouracil or gemcitabine as a radiosensitizer in the adjuvant setting.
2. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form.
3. Pregnant or breast feeding females (lactating females must agree not to breast feed while taking lenalidomide).
4. Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
5. Surgery or radiation therapy within 14 days of study enrollment as outlined below.

   * Surgery within 14 days of the start of study (patients must have recovered from effects of surgery; 7 days may be considered for minor procedures).
   * Palliative radiation therapy within 14 days of the start of study. The radiation therapy may not be to the only site of measurable disease.
6. Known brain or leptomeningeal disease (CT scan or MRI of the brain required only in case of clinical suspicion of central nervous system involvement).
7. Neuropathy of ≥ grade 2.
8. Known chronic infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Infante, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (9):
- United States (9):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide/Gemcitabine: The study began with a lead-in portion to confirm the tolerability of lenalidomide (25mg PO days 1-21) in combination with gemcitabine (1000mg/m2 IV days 1, 8, and 15). After completion of the lead-in phase, all subsequent patients received lenalidomide 25mg PO on days 1-21 and gemcitabine 1000mg/m2 IV days 1, 8, and 15 of 28-day treatment cycles. Patients were instructed to take lenalidomide at approximately the same time each morning. Patients were permitted to continue treatment until disease progression or intolerable toxicity occurred.
Period: Overall Study
Arm/Group | Lenalidomide/Gemcitabine
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide/Gemcitabine
Number analyzed (Participants) | 72
Age Continuous [Median (Full Range); unit: years] | 64 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Six-Month Overall Survival (OS) Probability, the Percentage of Patients Estimated to be Alive Six Months After Beginning Protocol Treatment
Description: The percentage of patients who were alive 6 months after beginning treatment
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide/Gemcitabine
Number analyzed (Participants) | 72
percentage of participants | 37 [26 to 48]

2. Secondary Outcome: Progression Free Survival (PFS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease
Description: The length of time, in months, that patients were alive from their first date of protocol treatment until worsening of their disease
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide/Gemcitabine
Number analyzed (Participants) | 72
months | 2.3 [1.9 to 3.5]

3. Secondary Outcome: Overall Survival (OS), the Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Description: Length of time, in months, that patients were alive from their first date of protocol treatment until death
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide/Gemcitabine
Number analyzed (Participants) | 56
months | 4.7 [3.4 to 5.7]

ADVERSE EVENTS:
Arm/Group | Lenalidomide/Gemcitabine
Serious Adverse Events (participants affected / at risk) | 8/72
Other Adverse Events (participants affected / at risk) | 71/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide/Gemcitabine (N=72)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Infection - Sepsis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 3 (3)
Perforation, GI (Gastrointestinal disorders) | 1 (1)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 (2)
Supraventricular arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1)
Splenic Abscess (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide/Gemcitabine (N=72)
Alkaline phosphatase (Metabolism and nutrition disorders) | 10 (16)
ALT (Metabolism and nutrition disorders) | 14 (17)
Neutrophils (Blood and lymphatic system disorders) | 27 (91)
Anorexia (Gastrointestinal disorders) | 27 (37)
Anxiety (Psychiatric disorders) | 6 (8)
Chills (Nervous system disorders) | 7 (7)
Confusion (Psychiatric disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 25 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Dehydration (Gastrointestinal disorders) | 13 (25)
Depression (Psychiatric disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 21 (32)
Dizziness (Nervous system disorders) | 11 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (20)
Edema - limb (Blood and lymphatic system disorders) | 23 (32)
Fatigue (General disorders) | 46 (88)
Fever (General disorders) | 11 (18)
Hemoglobin (Blood and lymphatic system disorders) | 45 (111)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 9 (15)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (12)
Hypokalemia (Metabolism and nutrition disorders) | 12 (24)
Hyponatremia (Metabolism and nutrition disorders) | 9 (14)
Hypotension (Cardiac disorders) | 8 (9)
Infection - urinary tract (Infections and infestations) | 4 (4)
Insomnia (Nervous system disorders) | 6 (9)
Jaundice (Hepatobiliary disorders) | 5 (7)
Leukocytes (Blood and lymphatic system disorders) | 24 (77)
Nausea (Gastrointestinal disorders) | 33 (51)
Neuropathy - sensory (Nervous system disorders) | 8 (10)
Pain - abdomen (General disorders) | 30 (46)
Pain - back (General disorders) | 13 (15)
Pain - chest (General disorders) | 12 (21)
Pain - headache (General disorders) | 7 (9)
Pain - limb (General disorders) | 9 (14)
Pain - stomach (General disorders) | 5 (6)
Platelets (Blood and lymphatic system disorders) | 41 (147)
Pruritis (Skin and subcutaneous tissue disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 22 (33)
Taste alteration (Gastrointestinal disorders) | 6 (7)
Thrombus/thrombosis/embolism (Vascular disorders) | 20 (27)
Tremor (Nervous system disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 15 (21)
Weakness (General disorders) | 11 (21)
Weight loss (General disorders) | 11 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.